CLINICAL TRIAL: NCT00883688
Title: A Phase II Study of Bevacizumab and Lapatinib in Children With Recurrent or Refractory Ependymoma
Brief Title: Bevacizumab and Lapatinib in Children With Recurrent or Refractory Ependymoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: CERN Foundation - Collaborative Ependymoma Research Network (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CERN08-01; NCI-2012-02129 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2009-04-17; First posted 2009-04-20 (Estimated); Results first posted 2020-08-26 (Actual); Last update posted 2020-08-26 (Actual); Status verified 2020-08

CONDITIONS: Brain Cancer; Pediatric Cancers
Keywords: Brain Tumor; Recurrent Ependymoma; Refractory Ependymoma; Intracranial ependymoma; Ependymoblastoma; Subependymoma; Myxopapillary; Clear cell; Anaplastic; Bevacizumab; Avastin; Anti-VEGF Monoclonal Antibody; rhuMAb-VEGF; Lapatinib; Tykerb; GW572016
MeSH Terms: conditions — Brain Neoplasms; Ependymoma; Neuroectodermal Tumors, Primitive; Glioma, Subependymal | interventions — Bevacizumab; Lapatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bevacizumab + Lapatinib (Experimental): Bevacizumab 10 mg/kg given by vein over 90 minutes for first injection (30-60 minutes for subsequent doses) every 2 weeks while on study (2 times during each 4-week "study cycle"). Lapatinib Pills of 700 mg/m^2/dose given orally 2 times each day.
  Interventions: Drug: Bevacizumab; Drug: Lapatinib

INTERVENTIONS:
Drug: Bevacizumab — 10 mg/kg given by vein over 90 minutes for first injection (30-60 minutes for subsequent doses) every 2 weeks while on study (2 times during each 4-week "study cycle").
  Other Names: Avastin; Anti-VEGF monoclonal antibody; rhuMAb-VEGF
Drug: Lapatinib — Pills of 700 mg/m^2/dose given orally 2 times each day.
  Other Names: Tykerb; GW572016

SUMMARY:
The goal of this clinical research study is to learn if the combination of Avastin (bevacizumab) and Tykerb (lapatinib) can help to control ependymoma in pediatric patients. The safety of this drug combination will also be studied.

DETAILED DESCRIPTION:
The Study Drugs:

Bevacizumab is designed to block the growth of blood vessels that supply nutrients necessary for tumor growth. This may prevent and/or slow down the growth of cancer cells.

Lapatinib is designed to prevent or slow down the growth of cancer cells by blocking proteins inside the cancer cells.

Study Drug Administration:

If you are found to be eligible to take part in this study, you will receive bevacizumab every 2 weeks while you are on study (2 times during each 4-week "study cycle"). The first time you receive the drug, it will be given by vein over 90 minutes. If this dose is well tolerated, you may receive future doses over 30 minutes.

You will take pills of lapatinib 2 times each day while you are on study. The pills should be taken at about the same time each day. You should not eat or drink anything except water for 1 hour before or 1 hour after you take the pills. If you miss a dose, do not take extra pills the next day to try and make up for the missed dose. You should report any missed pills or any trouble you may have with taking the pills to your study doctor.

You will be given a patient diary in which you must record what time you take lapatinib each time.

Study Visits:

At all study visits, you will be asked about any other drugs that you may be taking and about any side effects that you may be experiencing.

During Cycle 1 the following tests and procedures will be performed at least 1 time each week:

* You will have a physical exam, including measurement of your vital signs.
* Your performance status will be recorded.

Two (2) times each week during Cycle 1, blood (about 2-3 teaspoons) will be drawn for routine tests.

At the end of Cycle 1, urine will be collected for routine tests.

On Days 1 and 15 of Cycle 2, the following tests and procedures will be performed:

* You will have a physical exam, including measurement of your vital signs.
* Your performance status will be recorded.
* Blood (about 2-3 teaspoons) will be drawn for routine tests.

At the end of Cycle 2, you will have an MRI scan of your head to check the status of the disease. If your doctor thinks it is needed, you will also have an MRI of your spine and a spinal tap to check your cerebrospinal fluid (CSF) for presence of disease.

On Day 1 of Cycle 3 and beyond, the following tests and procedures will be performed:

* You will have a physical exam, including measurement of your vital signs.
* Your performance status will be recorded.
* Blood (about 2-3 teaspoons) and urine will be collected for routine tests.

Every 8 weeks, starting with the end of Cycle 4, while you are on study, the following tests and procedures will be performed:

* You will have an MRI scan of the brain to check the status of the disease.
* If your doctor thinks it is needed, you will have an MRI scan of the spine to check the status of the disease.
* If your doctor thinks it is needed, you will have a spinal tap to check your CSF for the presence of disease.

Every 12 weeks while you are on study, the following tests and procedures will be performed to check for possible side effects:

* You will have an echocardiogram or a multiple gated acquisition scan (MUGA) (if the study doctor thinks it is necessary) to test your heart function.
* You will have an x-ray of your right knee.
* If your doctor thinks it is needed, you will have an MRI scan of both knees.

Length of Study:

You will be on study for up to 2 years. You will be taken off study if the disease gets worse, if you experience intolerable side effects, or if the doctor thinks it is in your best interest.

End-of-Treatment Visit:

After you have finished receiving the study drugs, the following tests and procedures will be performed:

* You will have a physical exam, including measurement of your vital signs.
* You will be asked about any other drugs that you may be taking and about any side effects that you may be experiencing.
* Your performance status will be recorded.
* Blood (about 2-3 teaspoons) will be collected for routine tests.
* You will have an echocardiogram or a MUGA scan (if the study doctor thinks it is necessary) to test your heart function.
* You will have an x-ray of your right knee.
* You will have MRI scans of the brain and spine to check the status of the disease.
* If your doctor thinks it is needed, you will have a spinal tap to check the status of the disease.

Long-Term Follow-up:

You will have a follow-up visit 30 days after you have finished receiving the study drugs. The following tests and procedures will be performed:

* You will have a physical exam, including measurement of your vital signs.
* You will be asked about any other drugs that you may be taking and about any side effects that you may be experiencing.
* Your performance status will be recorded.
* Blood (about 2-3 teaspoons) will be collected for routine tests.

This is an investigational study. Bevacizumab is FDA approved and commercially available for the treatment of colon, rectum, lung and certain types of breast cancer. Lapatinib is FDA approved and commercially available for the treatment of certain types of breast cancer. The use of this drug combination in ependymomas in pediatric patients is investigational.

Up to 40 patients will take part in this multicenter study. Up to 6 patients will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Age: Patient must be < or = 21 years of age.
2. Tumor: Patients must have recurrent or refractory intracranial ependymoma (including myxopapillary, clear cell, papillary, tanycytic, and anaplastic ependymoma) or subependymoma. Patients with primary diagnosis of intracranial ependymoma with spinal cord metastases or relapse are eligible. The diagnosis must be confirmed by the CERN enrolling site's pathologist on tissue from either the initial presentation or time of recurrence prior to registration. For central pathology review and trial biological studies, submission of a paraffin block with tumor measuring at least 1 cm x 1 cm in area is preferred, but 15 x 5micro m unstained sections on slides may be provided by the referring laboratory instead. Tissue must be submitted within 60 days after enrollment for central processing and analysis.
3. Patients must have measureable disease which is defined as at least one measurable lesion that can be accurately measured in 2 planes. Diffuse leptomeningeal involvement ("sugar coating") that does not allow measurement of at least one lesion in 2 planes will not be considered measurable disease.
4. Patients may have had any number of prior treatment regimens (including biologic) before or after radiotherapy. Patients may not have previously been treated with Bevacizumab or Lapatinib. Gliadel wafers must be approved by CERN PI (Project Leader, Co-Leader and Protocol PI).
5. Neurological Deficits: Patients with neurological deficits should have deficits that are stable or improving for a minimum of 1 week prior to registration.
6. Performance Score: Karnofsky Performance Scale (KPS for > 16 years of age) or Lansky Performance Score (LPS for < or = 16 years of age) > or = 50 assessed within 2 weeks prior to registration.
7. Evidence of recovery from any prior chemotherapy. No myelosuppressive anticancer chemotherapy or biological therapy within 3 weeks (6 weeks if a nitrosourea or mitomycin C agent) prior to registration.
8. Prior/Concurrent Therapy: external beam radiation therapy (XRT): Patients must have had prior radiation therapy for treatment of their ependymoma. XRT must be > or = 3 months prior to registration for craniospinal irradiation (> or = 18 Gy); > or = 4 weeks for local radiation to primary tumor; and > or = 2 weeks prior to registration for focal irradiation to symptomatic metastatic sites.
9. Prior/Concurrent Therapy: Bone Marrow Transplant: > or = 3 months prior to registration for autologous bone marrow/stem cell transplant.
10. Prior/Concurrent Therapy: Anti-convulsants: Patients with seizure disorder may be enrolled if well controlled. Patients receiving enzyme-inducing anticonvulsants are not eligible for this study. Patients must be off EIACD for at least 2 weeks prior to registration.
11. Prior/Concurrent Therapy: Corticosteroids: Patients who are receiving corticosteroids must be on a stable or decreasing dose for at least 1 week prior to registration.
12. Prior/Concurrent Therapy: Growth Factors: Off all colony forming growth factor(s) > or = 2 weeks prior to registration (G-CSF, GM-CSF, Erythropoietin).
13. Patients must not have received: cytochrome P450 3A4 (CYP3A4) inhibitors within seven (7) days prior to registration on protocol and for the duration of the study. However, amiodarone, another CYP3A4 inhibitor, should have been discontinued 6 months prior to registration and for the duration of the study.
14. Patient must not have received: CYP3A4 inducers within fourteen (14) days prior to registration and for the duration of the study.
15. Patient must not have received: Cimetidine within 48 hours prior and for the duration of the study.
16. The following laboratory values must be assessed within 7 days prior to registration and must be repeated if initial labs were done greater than (>seven) (7) calendar days prior to the start of therapy. Organ Function: Must have adequate organ function and marrow function as defined by the following parameters: Bone Marrow: Absolute neutrophil count >or =1000microliter, Platelets > or = 100,000 microliter (transfusion independent), Hemoglobin >or =8.0 g/dL. Renal: Serum creatinine <or = 1.5 times upper limit of institutional for age or glomerular filtration rate (GFR)>or = 70ml/min/1.73m2 Hepatic: Total bilirubin < or = 1.5 times upper limit of normal for age: serum glutamate pyruvate transaminase (SGPT) (ALT)<2.5x institutional upper limit of normal for age and albumin > or = 2g/dL. No overt renal, hepatic, cardiac or pulmonary disease.
17. No overt renal, hepatic, cardiac or pulmonary disease.
18. Adequate cardiac function, assessed within 2 weeks prior to registration, defined as: shortening fraction of > or = 27% by echocardiogram, or ejection fracture (LVEF) > or = 50% by gated radionucleotide study.
19. Adequate pulmonary function, assessed within 2 weeks prior to registration, defined as: no evidence of dyspnea at rest, no exercise intolerance, and a pulse oximetry > 94% if there is clinical indication for determination.
20. Signed informed consent according to institutional guidelines must be obtained.
21. Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately and will be removed from the study.
22. Patient must begin therapy within 7 calendar days of registration.

Exclusion Criteria:

1. Patients may not have previously been treated with Bevacizumab or Lapatinib.
2. Patients with any significant medical illnesses that, in the investigator's opinion, cannot be adequately controlled with appropriate therapy or would compromise the patient's ability to tolerate this therapy.
3. Patients with any disease that would obscure toxicity or dangerously alter drug metabolism.
4. Patients receiving any other anticancer or experimental drug therapy.
5. Patients with uncontrolled infection.
6. Patients on enzyme inducing anticonvulsants.
7. Patients with > / = Grade 2 uncontrolled hypertension.
8. History of a stroke, myocardial infarction, or unstable angina in the previous 6 months.
9. Evidence of a bleeding diathesis, coagulopathy or PT international normalized ratio (INR)>1.5.
10. Patients who require the use of therapeutic anti-coagulation: except as required to maintain patency of preexisting permanent vascular catheter.
11. Pre-existing coagulopathy or thrombosis: Patients must not have been previously diagnosed with a deep venous or arterial thrombosis (including pulmonary embolism), and must not have a known thrombophilic condition.
12. Patients must have recovered from any surgical procedure before enrolling on this study.
13. History of an abdominal fistula, GI perforation, or intra-abdominal abscess within previous 6 months.
14. A serious, non healing wound, ulcer, or bone fracture.
15. Evidence of a new intracranial or intratumoral hemorrhage that is larger than a punctuate size on baseline MRI obtained within 14 days prior to study registration.
16. If there is proteinuria present on dipstick, patients must have a 24 hour urine collection. Patients are excluded if they have >500 mg protein on 24 hour urine collection.
17. Pregnancy: Females of childbearing potential must have negative serum or urine pregnancy test within 7 days prior to study entry. The effects of lapatinib on the developing human fetus are unknown. However, bevacizumab is known to be teratogenic and detrimental to fetal development and endometrial proliferation, thereby having a negative effect on fertility.
18. Breastfeeding: Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with lapatinib of bevacizumab, breastfeeding should be discontinued if the mother is treated on this study.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2009-07; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael E. Rytting, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (6):
- United States (6):
  - Stanford University Medical Center, Stanford, California
  - Children's Memorial Hospital, Chicago, Illinois
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - University of Texas MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: July 23, 2009 to April 3, 2013. All recruitment done in medical clinics.
Groups:
- Bevacizumab + Lapatinib: Bevacizumab 10 mg/kg intravenous over 90 minutes for first injection (30-60 minutes for subsequent doses) every 2 weeks while on study (2 times during each 4-week "study cycle"). Lapatinib 700 mg/m^2/dose given orally 2 times each day.
Period: Overall Study
Arm/Group | Bevacizumab + Lapatinib
Started | 24
Completed | 22
Not Completed | 2
Not completed — Ineligible | 2

BASELINE CHARACTERISTICS:
Arm/Group | Bevacizumab + Lapatinib
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 24
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 17
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: Objective response rate defined as number of participants out of total participants with complete response plus partial response (CR+PR) sustained for at least four weeks. Complete Response (CR) - Complete disappearance on magnetic resonance imaging (MRI) of all enhancing tumor and mass effect, on a stable or decreasing dose of corticosteroids (or receiving only adrenal replacement doses), accompanied by a stable or improving neurologic examination and must be sustained for at least 4 weeks. If cerebrospinal fluid (CSF) for presence of disease was positive it must become negative. Partial Response (PR) - Greater than or equal to 50% reduction in tumor size by bi-dimensional measurement on a stable or decreasing dose of corticosteroids, accompanied by stable or improving neurological examination and must be sustained for at least 4 weeks.
Time Frame: 4 weeks following treatment, repeat assessments up to one year.
Population: Of the total, 22 participants were eligible and only 20 evaluable for response.
Measure: Number; unit: Percentage of Participants
Arm/Group | Bevacizumab + Lapatinib
Number analyzed (Participants) | 20
Percentage of Participants | 0

ADVERSE EVENTS:
Time Frame: Adverse event collection through 8 week treatment and may continue for up to 26 courses (2 years).
Arm/Group | Bevacizumab + Lapatinib
Serious Adverse Events (participants affected / at risk) | 11/24
Other Adverse Events (participants affected / at risk) | 24/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bevacizumab + Lapatinib (N=24)
Increase serum glutamic pyruvic transaminase (ALT, SGPT) (Investigations) | 3 (4)
Apnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Increase serum glutamic oxaloacetic transaminase (AST, SGOT) (Investigations) | 1 (1)
Increase creatine phosphokinase (CPK ) (Investigations) | 1 (1)
Pustular Rash/Scalp (Skin and subcutaneous tissue disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) — Fever of unknown origin without clinically or microbiologically documented infection (ANC <1.0 x 10^9/L, fever >=38.5 degrees C)
High gamma-Glutamyl transpeptidase (GGT) (Investigations) | 1 (1)
Hemorrhage, Central Nervous System (Nervous system disorders) | 1 (1)
Hemorrhage: Respiratory tract NOS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils : Abdomen NOS (Infections and infestations) | 1 (1)
Left ventricular systolic dysfunction (Cardiac disorders) | 1 (1)
Cranial Neuropathy CN IX Motor (Nervous system disorders) | 2 (2)
Gastrointestional Obstruction: Gallbladder (Hepatobiliary disorders) | 1 (1)
Abdomen Pain (Gastrointestinal disorders) | 1 (1)
Extremity Pain, Limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Somnolence/depressed level of consciousness (Nervous system disorders) | 1 (1)
Speech impairment (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bevacizumab + Lapatinib (N=24)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 3 (9)
Alkaline phosphatase (Investigations) | 2 (3)
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Allergy - Bumpy tongue (Immune system disorders) | 1 (1)
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 7 (16)
Anorexia (Metabolism and nutrition disorders) | 7 (9)
Apnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (2)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Investigations) | 7 (14)
Ataxia (incoordination) (Nervous system disorders) | 12 (14)
Hearing loss (Ear and labyrinth disorders) | 1 (1)
Bicarbonate, serum-low (Investigations) | 1 (1)
Bilirubin (hyperbilirubinemia) (Investigations) | 4 (5)
Bronchospasm, wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 1 (1)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 3 (13)
Coagulation: Activated partial thromboplastin time (aPTT or APTT) (Investigations) | 1 (2)
Cognitive disturbance (Nervous system disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 6 (9)
Constitutional Symptoms (General disorders) | 3 (3) — Changes in appearance, voice, appetite
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3)
CPK (creatine phosphokinase) increase (Investigations) | 1 (1)
Creatinine Increases (Investigations) | 1 (4)
Cushingoid appearance (e.g., moon face, buffalo hump, centripetal obesity, cutaneous striae) (Endocrine disorders) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 3 (3)
Sores & pustules (Skin and subcutaneous tissue disorders) | 5 (5)
Diarrhea (Gastrointestinal disorders) | 18 (44)
Dizziness (Nervous system disorders) | 2 (2)
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 1 (1)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Edema: limb (General disorders) | 1 (1)
Extremity-lower (gait/walking) (General disorders) | 1 (1)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 14 (17)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) — Fever of unknown origin without clinically or microbiologically documented infection (ANC <1.0 x 10^9/L, fever >=38.5 degrees C)
Fever (General disorders) | 2 (2) — In absence of neutropenia, where neutropenia defined as ANC <1.0 x 10^9/L
Flatulence (Gastrointestinal disorders) | 1 (1)
Gastrointestinal - Other (Blood in stool, gas) (Gastrointestinal disorders) | 1 (4)
GGT (gamma-Glutamyl transpeptidase) (Investigations) | 1 (2)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 1 (4)
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 1 (2)
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 4 (4)
Hearing: patients with/without baseline audiogram and enrolled in a monitoring program (Ear and labyrinth disorders) | 1 (1)
Heartburn/dyspepsia (Gastrointestinal disorders) | 1 (1)
Hemoglobin Change (Investigations) | 3 (7)
Hemorrhage, CNS (Nervous system disorders) | 1 (1)
Hemorrhage, pulmonary/upper respiratory : Nose (Respiratory, thoracic and mediastinal disorders) | 4 (9)
Hemorrhage, pulmonary/upper respiratory : Respiratory tract NOS (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Hypertension (Vascular disorders) | 3 (3)
Hypotension (Vascular disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Incontinence, urinary (Renal and urinary disorders) | 2 (2)
Infection - Other (Specify, Upper Respiratory) (Infections and infestations) | 2 (4)
Infection with normal ANC, Grade 1/2 neutrophils (Infections and infestations) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils : Abdomen NOS (Infections and infestations) | 1 (1)
Infection normal ANC or Grade 1 or 2 neutrophils: Foreign body (Infections and infestations) | 2 (2) — Foreign body (e.g., graft, implant, prosthesis, stent)
Infection with normal ANC or Grade 1 or 2 neutrophils : Trachea (Infections and infestations) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils : Urinary tract NOS (Infections and infestations) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils : Vagina (Infections and infestations) | 1 (1)
Infection with unknown ANC : Lung (pneumonia) (Infections and infestations) | 1 (1)
Infection with unknown ANC : Urinary tract NOS (Infections and infestations) | 1 (1)
INR (International Normalized Ratio of prothrombin time) (Investigations) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2)
Laryngeal nerve dysfunction (Nervous system disorders) | 1 (1)
Left ventricular systolic dysfunction (Cardiac disorders) | 1 (1)
Lumbar spine-range of motion (Musculoskeletal and connective tissue disorders) | 1 (1)
Lymphatics - Other (Specify, swollen hands) (Vascular disorders) | 1 (1)
Lymphopenia (Vascular disorders) | 3 (6)
Magnesium, serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 1 (1)
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 2 (2)
Metabolic/Laboratory - Other (Specify, phosphorus increase) (Investigations) | 1 (1)
Mood alteration : Anxiety (Psychiatric disorders) | 2 (2)
Mood alteration : Depression (Psychiatric disorders) | 1 (1)
Mucositis/stomatitis (clinical exam) : Oral cavity (Gastrointestinal disorders) | 1 (1)
Mucositis/stomatitis (functional/symptomatic) : Oral cavity (Gastrointestinal disorders) | 3 (3)
Muscle weakness, generalized or specific area (not due to neuropathy) : Extremity-lower (Musculoskeletal and connective tissue disorders) | 2 (2)
Muscle weakness, generalized or specific area (not due to neuropathy) : Left-sided (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness, generalized or specific area (not due to neuropathy) : Right-sided (Musculoskeletal and connective tissue disorders) | 1 (1)
Weakness, limp (Musculoskeletal and connective tissue disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 7 (9)
Central Nervous System (CNS) affectation (Nervous system disorders) | 5 (5)
Cranial Neuropathy: CN IX Motor-pharynx (Nervous system disorders) | 4 (4) — Sensory-ear, pharynx, tongue
Cranial Neuropathy: CN VI Lateral deviation of eye (Nervous system disorders) | 2 (2)
Cranial Neuropathy: CN VII Motor-face (Nervous system disorders) | 3 (3) — Sensory-taste
Cranial Neuropathy: CN X Motor-palate (Nervous system disorders) | 1 (1) — pharynx, larynx
Cranial Neuropathy: CN XII Motor-tongue (Nervous system disorders) | 2 (2)
Motor Neuropathy (Nervous system disorders) | 3 (3)
Sensory Neuropathy (Nervous system disorders) | 3 (3)
Nystagmus (Nervous system disorders) | 6 (7)
Obesity (Metabolism and nutrition disorders) | 1 (1)
Obstruction, GI : Gallbladder (Hepatobiliary disorders) | 1 (1)
Ptosis, dry eyes (Eye disorders) | 3 (4)
Ophthalmoplegia/diplopia (double vision) (Eye disorders) | 4 (4)
Otitis, external ear (non-infectious) (Ear and labyrinth disorders) | 1 (2)
Knee Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain - Neck (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain - Thigh (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain : Abdomen NOS (Gastrointestinal disorders) | 7 (7)
Pain : Back (Musculoskeletal and connective tissue disorders) | 2 (3)
Pain : External ear (Ear and labyrinth disorders) | 1 (1)
Pain : Extremity-limb (Musculoskeletal and connective tissue disorders) | 3 (3)
Pain : Head/headache (Nervous system disorders) | 7 (12)
Pain : Muscle (Musculoskeletal and connective tissue disorders) | 3 (3)
Pain : Oral cavity (Gastrointestinal disorders) | 1 (1)
Pain : Stomach (Gastrointestinal disorders) | 2 (2)
Pain : Throat/pharynx/larynx (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 6 (8)
Platelets low (Blood and lymphatic system disorders) | 1 (2)
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 1 (1)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 5 (9)
Prolonged intubation after pulmonary resection (>24 hrs after surgery) (Investigations) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 2 (5)
Partial Thromboplastin Time (PTT) outside normal (Investigations) | 1 (1)
Respiratory arrest/choking, congestion, tachypnea (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 12 (23)
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 3 (3)
Renal failure (Renal and urinary disorders) | 1 (1)
Renal/Genitourinary - Other (urination issues) (Renal and urinary disorders) | 1 (1)
Seizure (Nervous system disorders) | 2 (2)
Sodium, serum-high (hypernatremia) (Metabolism and nutrition disorders) | 1 (1)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 2 (3)
Somnolence/depressed level of consciousness (Nervous system disorders) | 1 (1)
Speech impairment (e.g., dysphasia or aphasia) (Nervous system disorders) | 3 (3)
Striae (Skin and subcutaneous tissue disorders) | 1 (1)
Thyroid function, low (hypothyroidism) (Endocrine disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Triglyceride, serum-high (hypertriglyceridemia) (Metabolism and nutrition disorders) | 1 (1)
Urinary retention (including neurogenic bladder) (Renal and urinary disorders) | 2 (2)
Valvular heart disease (Cardiac disorders) | 1 (1)
Vision-blurred vision (Eye disorders) | 1 (1)
Voice changes/dysarthria (e.g., hoarseness, loss or alteration in voice, laryngitis) (Immune system disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 8 (10)
Weight loss (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No